CLINICAL TRIAL: NCT01023542
Title: A 3-Armed Prospective Randomized Controlled, Open-Labeled Phase II Trial to Evaluate Late Introduction of Cyclosporine or Everolimus Versus a 5-day Delay of Cyclosporine in Combination With MMF in Liver Transplant Recipients With MELD-Scores≥25
Brief Title: CNI-free "Bottom"-up Immunosuppression in Patients Undergoing Liver Transplantation
Acronym: BUILT_01
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Regensburg (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Regensburg University, Regensburg University Hospital, Department of Surgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BUILT_01
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Renal Impairment; Liver Transplantation; Everolimus
Keywords: renal impairment; MELD>25; Liver transplantation; CNI-free; Bottom-Up; Everolimus
MeSH Terms: conditions — Renal Insufficiency | interventions — cni protein, Drosophila

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Basiliximab 20 mg day 0 and 4 + MMF 2x1 g i.v./d from day 0 (will be switched to oral administration after 1 week) + low level cyclosporine [start at day 5 after OLT, trough-level 100-150 ng/mL (CsA)] + low-level steroids 1 mg/kg KG/d from day 0, elimination by month 6 after LTx.
  Interventions: Drug: delayed, low-dose CNI
- 2 (Active Comparator): Basiliximab 20 mg Tag 0 and 4 + MMF 2x1 g i.v./d from day 0 (will be switched to oral administration after 1 week) + low-level steroids 1 mg/kg KG/d from day 0, elimination by month 6 after LTx + low-level cyclosporine (start within 30 days after LTx; trough level 100-150ng/mL (CsA).
  Interventions: Drug: BU-CNI
- 3 (Experimental): Basiliximab 20 mg Tag 0 and 4 + MMF 2x1 g i.v./d from day 0 (will be switched to oral administration after 1 week) + low-level steroids 1 mg/kg KG/d from day 0, elimination by month 6 after LTx + everolimus (start within 30 days after LTx; trough-level 6-10 ng/mL).
  Interventions: Drug: BU-Everolimus

INTERVENTIONS:
Drug: delayed, low-dose CNI — immunosuppression
  Arms: 1
Drug: BU-CNI — Immunosuppression
  Arms: 2
Drug: BU-Everolimus — Immunosuppression
  Arms: 3

SUMMARY:
The primary objective of the trial is to evaluate efficacy and safety of delayed introduction (up to 30 days post-transplantation in patients without signs of acute rejection that had received an aIL-2 induction and MMF) of either cyclosporine or everolimus versus a 5-day delay of cyclosporine in combination with MMF.

DETAILED DESCRIPTION:
The risk of developing chronic renal failure after liver transplantation (LT) in the pre-MELD era was approximately 20% after 5 years, associated with the use of CNI and a 4-fold increased mortality risk. Besides pre-transplant factors associated with end-stage hepatic disease that influence renal function (hepatorenal syndrome [HRS]), there are major risk factors associated with early post-transplant renal impairment: preexisting diabetes mellitus, time on the waiting list with end-stage hepatic disease, requirement for blood products, liver allograft dysfunction, HCV-infection and toxicity of Calcineurin-inhibitors (CNI) (1-8). The introduction of the MELD-based allocation system in the Eurotransplant area in December 2006 led to an increase of the proportion of liver transplant recipients with renal dysfunction before and at the time of liver transplantation (LT), since creatinine became a key component for the allocation of liver allografts (9). Data from 2 recent publications indicate an incidence of pre-transplant renal impairment with an eGFR ≤ 60ml/min. of approximately 50%. Renal impairment and MELD-scores ≥ 24 as well as the requirement for renal replacement therapy before LT result in a significantly unfavorable outcome after LT (10,11). An additional problem in this specific patient group (impaired renal function at the time of LT and MELD-scores ≥ 25), is a high risk for developing infectious complications (12). Studies indicate that early infections are present in almost 85% of all patients, and become the most common cause of death early after transplantation. Notably, two-third of infections in liver transplant patients occur within the first 3 months after transplantation with a very high percentage (67%) of severe infections (13,14). In general, the inflammatory response associated with infection is impaired by immunosuppressive drugs. This disturbed regulation increases the susceptibility for a broad range of normal and of opportunistic infections (15). Therefore, patients with high lab-MELD scores hypothetically should require a rather low amount of immunosuppressive (IS) drugs during the first days to weeks after transplantation, while they are in a state of SIRS (systemic inflammatory response syndrome)-like state (16,17). In Regensburg a collective of 30 patients with renal impairment (creatinine of 1.5 g/dL or higher and/or eGFR of 50 ml/min or lower) at the time point of LT, or on day 1 after LT, was treated with either standard CNI + MMF + basiliximab + steroids (control-arm; group 2) or with a CNI-free protocol consisting of MMF + basiliximab + steroids (treatment-arm; group 1). Baseline renal function was similar: serum creatinine (SCr) median 1.8 mg/dL (1.5 to 4.0 mg/dL) (group A) vs. 2.4 mg/dL (1.5 to 4.0 mg/dL) (group B) [p=0.24]. Results from our retrospective case-control study show that the cumulative requirement for renal replacement therapy was significantly lower in group B (p=0.032). Ten of 15 patients received additional immunosuppression (4 CNI and 6 mTOR inhibitor) beyond day 30. By month 6 (1.3 mg/dL vs. 1.1 mg/dL) and month 12 (1.6 mg/dL vs. 1.2 mg/dL), group B patients showed significantly better SCr (and eGFR) values than group A (p=0.006). Rates of BPAR were similar, but pulmonary complications were higher in group A resulting in a significantly longer stay on ICU (9 vs. 21 days; p=0.04). The investigators concluded from this collective that CNI-free-"bottom-up" immunosuppression in severely ill patients with renal impairment prior to LT is feasible and may be an innovative approach to improve outcome (18). Based on these initial findings the investigators initiated a prospective uncontrolled two-step pilot-trial to investigate the safety and efficacy of CNI-free de novo "bottom-up" immunosuppression in patients undergoing LT with existing renal impairment (PATRON07-study, clinicaltrials.gov-identifier: NCT00604357) (19). In the first step of this pilot trial, nine patients were treated with MMF 2x1g i.v./day, including induction therapy with basiliximab 20 mg i.v. on days 0 and 4, and center-specific steroids; sirolimus was introduced into the regimen at least 10 days after LT. The primary endpoint was the incidence of steroid-resistant biopsy-proven acute rejections at 30 days after transplantation, as an early detector of safety and efficacy. Analysis of the first nine patients confirmed our findings in the retrospective analysis summarized in section 2.1. Only one biopsy proven acute rejection occurred. No patient lost their allograft, and no patient died within one year after LT. Renal function improved significantly from baseline to 30 days, and to 3 and 6 months after transplantation (p=0.004). At 3 and 6 months, 72% of all patients were still CNI-free. All side-effects observed were expected for treatment with mTOR-inhibitors. Although the median lab MELD-score at baseline was 29 (range: 10 to 40), and the initial Karnowsky-index was 20 (range: 10 to 80), patients recovered quite quickly and had a Karnowsky-index of 60 (range: 20 to 80) at day 30 and 80 (range: 50 to 100) at 3 months after LT. These findings indicate the feasibility of CNI-free de novo "bottom-up" IS without increased risk for acute rejection, graft-loss and mortality but a beneficial impact on short- and long-term renal function as independent risk-factor for long-term mortality after LT.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female liver transplant recipients of a primary liver transplant older than 18 years
2. Signed, written informed consent prior to randomization
3. MELD scores ≥25
4. Lack of relevant exclusion criteria

Exclusion Criteria:

1. Patients transplanted for autoimmune hepatitis
2. HIV positive patients
3. Patients with pre-transplant immunosuppressive treatment
4. Patients who are recipients of multiple solid organ or islet cell tissue transplants, or have previously received an organ or tissue transplant.
5. Patients with renal failure or CKD/ESRD who require renal replacement therapy for more than 2 weeks prior to transplantation.
6. Patients with signs of hepatic artery thrombosis.
7. Patients with a hepatic encephalopathy grade of Stadium II, III and IV (somnolence, sopor and loss of consciousness
8. Patients with a known hypersensitivity to the drugs used on study or their class, or to any of the excipients.
9. Patients who are recipients of ABO incompatible transplant grafts.
10. Patients with uncontrolled or therapy refractory hypercholesterolemia (>350 mg/dL; >9 mmol/L) or hypertriglyceridemia (>500 mg/dL; >8.5 mmol/L) at time of transplantation.
11. Patients with platelet count <50,000/mm3 at the time of randomization.
12. Patients with an absolute neutrophil count of <1,000/mm³ or white blood cell count of <2,000/mm³ at the time of randomization.
13. Patients with a creatinine/protein ratio indicating daily urinary protein excretion > 1 g/24h at time of randomization.
14. Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS (1) they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m, or (2) have past 6 weeks from surgical bilateral oophorectomy with or without hysterectomy or (3) are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), copper coated IUD and double-barrier methods ( any double combination of male or female condom with spermicidal gel, diaphragm, sponge, cervical cap). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. Reliable contraception should be maintained throughout the and for 3 months after study drug discontinuation.
15. Patients with any history of coagulopathy or medical condition requiring long-term anticoagulation which would preclude liver biopsy after transplantation.
16. Patients with a psychologic, familial, sociologic or geographic condition potentially hampering compliance with the study protocol and follow-up schedule.
17. Patients under guardianship (e.g. individuals who are not able to freely give their informed consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of the trial is renal function at 12 months measured by estimated GFR using abbreviated MDRD formula. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Andreas A Schnitzbauer, MD, Principal Investigator — Regensburg University Hospital, Department of Surgery; Hans J Schlitt, MD, Study Chair — Regensburg University Hospital Department of Surgery
Locations (1):
- Regensburg University Hospital, Regensburg, Bavaria, Germany